CLINICAL TRIAL: NCT02074033
Title: Determination of Errors in Prescription Antibiotics in Ventilator-associated Pneumonia in Unit of Intensive Care of Clinical Hospital of Federal University of Uberlandia - Brazil
Brief Title: Errors in Prescription Antibiotics in Ventilator-associated Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Ana Carolina Souza Oliveira, graduate student, Federal University of Uberlandia
Other Study IDs: 30121978
Record Dates: First submitted 2014-02-23; First posted 2014-02-28 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: No samples will be retained for the study
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- antibiotics for pneumonia: We will be examined whether the antibiotic prescribed following the orientation of literature, considering the dose, interval between doses, dose adjustment for renal failure infusion time, treatment time and conduct after the culture results (deescalation, escalation or maintenance of antimicrobial initially prescribed )

SUMMARY:
The infection is a major risk to hospitalized patients, especially those admitted to the Intensive Care Unit (ICU) and an unfavorable factor in the outcome of critically ill patients, increasing costs and prolonging hospitalization hospitalar. The ventilator-associated pneumonia (PAV) is considered the most prevalent nosocomial infection in the ICU, occurring in 9% to 68% of patients with prosthetic ventilatória.Due to the high rate of PAV and mortality related to it, is very important both prescription and administration of antibiotics correctly, as deescalation or escalation according the result of cultures.Therefore, the objectives of this study is assess if whether the antibiotic prescribed of ventilator-associated pneumonia following the orientation of literature. Will also be assessed the rate of PAV in patients critically ill adults, the main microorganisms responsible by PAV and determining antimicrobial susceptibility.

DETAILED DESCRIPTION:
In patients who had a diagnosis of ventilator-associated pneumonia by asssistente physician will be assessed initially prescribed antibiotics empirically and what conduct adopted after culture results.

We will be examined whether the antibiotic prescribed following the orientation of literature, considering the dose, interval between doses, dose adjustment for renal failure infusion time, treatment time and conduct after the culture results (deescalation, escalation or maintenance of antimicrobial initially prescribed ) . The deescalation consists of discontinuing the use of antimicrobial or antibiotic change to another with lower coverage and spectrum is performed, escalation occurs when adding a new antibiotic or antibiotic to change the coverage of other larger spectrum after culture results .

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age;
* Having the diagnosis of ventilator-associated pneumonia.

Exclusion Criteria:

* Be under 18 years of age;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is a retrospective study to evaluate the use of antibiotics in the ventilator-associated pneumonia (PAV) in the Intensive Care Unit of the Adult Clinical Hospital of the Federal University of Uberlândia. The UnitAdult Intensive Care has complexity level III and consists of 30 beds.O number of statistically significant sample is 130 patients.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-04 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Determination of Errors in Prescription Antibiotics in Ventilator-associated Pneumonia in Unit of Intensive Care of Clinical Hospital of Federal University of Uberlandia - Brazil | six months

CONTACTS AND LOCATIONS:
Overall Officials: Ana Carolina Souza Oliveira, Principal Investigator — Federal University of Uberlandia; Denise Von Dollinger de Brito, Principal Investigator — Federal University of Uberlandia; Thúlio Marquez Cunha, Principal Investigator — Federal University of Uberlandia; Fabiola Alves Gomes, Principal Investigator — Federal University of Uberlandia
Locations (1):
- Ana Carolina Souza Oliveira, Uberlândia, Minas Gerais, Brazil

REFERENCES:
- See also: Guidelines for the Management of Adults with Hospital-acquired, Ventilator-associated, and Healthcare-associated Pneumonia. American Journal of Respiratory and Critical Care Medicine, New — http://www.ncbi.nlm.nih.gov/pubmed
- See also: ALVAREZ-LERMA, F. et al. Empiric broad-spectrum antibiotic therapy of nosocomial pneumonia in the intensive care unit: A prospective observational study. Crit Care, London, v.10, n.3, p.1-11, May 2006. — http://www.ncbi.nlm.nih.gov/pubmed
- See also: ANGUS, D.C.et al. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome and associa¬ted costs of care. Crit Care Med, New York, v.29, n.7, p.1303-1310, Jul 2001. — http://www.ncbi.nlm.nih.gov/pubmed
- See also: BURKE, J.P. Infection control- a problem for patient safety. N Engl J Med, Melbourn, v.348, n.7, p. 651-656, Feb 2003. — http://www.ncbi.nlm.nih.gov/pubmed
- See also: CAMARGO, L. F. A. et al. Ventilator associated pneumonia: comparison between quantitative and qualitative cultures of tracheal aspirates. Critical Care Medicine, New York, v.8, n.6, p. 422-430, Dec 2004. — http://www.ncbi.nlm.nih.gov/pubmed
- See also: EACHEMPATI, S.R. et al. Does de-escalation of antibiotic therapy for ventilator-associated pneumonia affect the likelihood of recurrent pneumonia or mortality in critically ill surgical patients? J Trauma, Baltimore, v.66, n.5, p.1343-1348, May 2009. — http://www.ncbi.nlm.nih.gov/pubmed
- See also: ERBAY, A., BODUR, H., AKINCI, E., ÇOLPAN, A. Evaluation of antibiotic use in intensive care units of a tertiary care hospital in Turkey. Journal of Hospital Infection, New York , v.59, p.53-61, Jan 2005. — http://www.ncbi.nlm.nih.gov/pubmed
- See also: GOMES SILVA, B.N. et al. De-escalation of antimicrobial treatment for adults with sepsis, severe sepsis or septic shock. Cochrane Database Syst Rev, Oxford,v.8, n.12, CD007934, Dec 2010. — http://www.ncbi.nlm.nih.gov/pubmed
- See also: HEENEN, S., JACOBS, F., VINCENT,J-P. Antibiotic strategies in severe nosocomial sepsis: Why do we not de-escalate more often? Crit Care Med, New York, v.40, n.5, p.1404-1409, May 2012 . — http://www.ncbi.nlm.nih.gov/pubmed
- See also: RELLO, J. et al. De-escalation therapy in ventilator associated pneumonia. Crit Care Med , New York, v.32, n.11, p.2183-2190, Nov 2004. — http://www.ncbi.nlm.nih.gov/pubmed
- See also: SAFDAR, N.; CRNICH, C.J.; MAKI, D.G. The Pathogenesis of Ventilator-Associated Pneumonia: Its Relevance to Developing Effective Strategies for Prevention. Respiratory Care, Philadelphia, v.50, n.6, p.725-739, Jun 2005. — http://www.ncbi.nlm.nih.gov/pubmed
- See also: WAELE, J.J.D.et al. De-escalation after empirical meropenem treatment in the intensive care unit: Fiction or reality? Journal of Critical Care, Orlando, v.25, n.4, p.641-646, Jan 2010. — http://www.ncbi.nlm.nih.gov/pubmed